CLINICAL TRIAL: NCT06298773
Title: SPATIAL PROFILE OF SUBPOPULATIONS OF CANCER AND IMMUNITARY CELLS IN SEVERAL SOLID TUMORS
Brief Title: Spatial Profile of Tumors
Acronym: PROST
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6127
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Spatial analysis of paraffin samples from solid tumors — The intervention involves the collection of tumour samples included in paraffin present in the pathological anatomy archive or requested to external archives for samples older than 2003 and the subsequent multiparametric spatial analysis of the main populations of the microenvironment tumor.

SUMMARY:
The research project focuses on analyzing the spatial organization of cells within various solid tumors, utilizing advanced technologies enabling in-depth multi-parametric analysis of tumor and immune cells. The primary objective is to understand the spatial distribution of cellular subpopulations within each type of tumor, while secondary objectives include correlating these data with clinical aspects and identifying potential therapeutic targets. The study involves 1000 patients with primary or metastatic tumors and spans a duration of 5 years, from 2024 to 2028. No experimental treatments are planned; rather, only spatial imaging analyses with multiple markers will be conducted. Data analysis involves descriptive statistical methods and hypothesis testing to generate hypotheses for subsequent studies. The analyses will be performed using SPSS® version 21.0 software for Windows®.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects aged 18 years
* primary or metastatic tumors Diagnosed by histology and/or radiological evidence, RNM, or endoscopic
* signature of informed consent
* substitute declaration to the consent form where applicable

Exclusion Criteria:

* previous unrelated tumour disease
* significant acute or chronic infections (HIV, HCV and HBV infections) and/or ongoing bacterial and viral infections
* active autoimmune disease
* pregnant or breastfeeding
* patients who do not sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be 1000 adult male and female patients with primary or metastatic neoplastic pathology of the following types of cancer: lung cancer, colon cancer, salivary gland cancer, hepatocarcinoma, sarcomas, osteosarcomas, breast cancer, glioblastoma, kidney cancer, pancreatic cancer, neck cancer.
  The patient samples that will be examined in the study are derived from biopsies that patients have been subjected to according to their treatment plan.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-05 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Spatial analysis of cancer cells | 7 days
  Spatial distribution analysis of the main cell subpopulations characterising the tumours studied.

SECONDARY OUTCOMES:
Comparison of clinical data | 1 day
  Correlation of spatial analysis data with patient clinical data
Identification of therapeutic targets | 4 weeks
  Identification of possible therapeutic targets of different subpopulations

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Sgambato, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, RM, Italy